CLINICAL TRIAL: NCT05907265
Title: Study of the Benefits of Immersive Virtual Reality Techniques on the Effects on Cognition in People With Cancer (OncoBRAIN)
Brief Title: Immersive Virtual Reality Techniques on the Effects on Cognition in People With Cancer
Acronym: OncoBRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Maite Garolera, Principal Investigator of the Brain, Cognition, and Behavior Research Group (C3-CST), Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-22-107-107
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cancer; Cognitive Impairment
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality group (Experimental): The intervention will be group-based, with 5 participants per group, and will consist of a total of 24 sessions of 60 minutes. These 24 sessions are organized over 12 weeks, 2 sessions per week. The sessions will consist of a group program of multimodal stimulation using immersive MK360 technology to train cognitive, emotional, and physical areas.
  Each session will have a different content, although they will follow the following outline:
  1. Welcome and awareness of the here and now.
  2. Mindfulness techniques
  3. Cognitive stimulation
  4. Physical activation
  5. Feedback and end of session.
  The visual material used for each session will be specific and adapted to the group.
  Interventions: Behavioral: Behavioral: ONCOBrain_ImmersiveVR
- Active Comparator: Active control program (Active Comparator): In paper or pdf format, patients in the active control group will receive guidelines for physical and cognitive stimulation to do autonomously at home. Patients in the active control group will receive guidelines for cognitive and physical stimulation and meditation exercises in paper or pdf format, to be done independently at home. They will be encouraged to do physical exercises, meditation, and cognitive activities two times a week.
  Interventions: Behavioral: Behavioral: Control_Condition

INTERVENTIONS:
Behavioral: Behavioral: ONCOBrain_ImmersiveVR — A multimodal and digitally-based cognitive training, physical exercise and mindfulness intervention delivered face to face and through 360MK Virtual Reality technology
  Arms: Immersive Virtual Reality group
Behavioral: Behavioral: Control_Condition — Traditional paper or pdf format multimodal intervention that will combine cognitive, mediation and physical activities.
  Arms: Active Comparator: Active control program

SUMMARY:
OncoBRAIN aims to assess the effect of an innovative immersive virtual reality-based (IVR) intervention that includes cognitive, physical activity and mindfulness exercises in people diagnosed with cancer and Chemotherapy-Related Cognitive Deficits (CRCD). The main objective of OncoBRAIN is to determine the benefits of RVI intervention on the cognitive, and emotional state and quality of life of people with cancer and CRQD. We hypothesize that in OncoBRAIN we will find improvements in people with cancer and CRCD who have received IVR stimulation compared to the control group with cancer and CRCD who have not received IVR stimulation. People in the experimental group will perform better than patients in the control group in cognition (episodic memory, executive function, attention, and information processing speed), show better emotional well-being and perceive a better quality of life at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

A. Over 18 years of age and under 65 years of age B. Diagnosis of cancer C. At least 4 weeks since the last chemotherapy treatment session D. Presence of cognitive complaints after chemotherapy treatment E. Level of primary education to be able to perform the cognitive tests. F. Consent to participate in the study

Exclusion Criteria:

A. Established diagnosis prior to cancer diagnosis of psychiatric, neurological, neurodevelopmental or systemic disorder causing cognitive deficits.

B. Motor or sensory impairments that preclude completion of the program. C. Undergoing chemotherapy treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in scores of global cognition | Before the intervention and 12 weeks later
  Global cognition was assessed with the Montreal Cognitive Assessment (MoCA) a screening tool designed to identify mild cognitive impairment (MCI) and other cognitive deficits. The MoCA takes around 10-15 minutes to complete and consists of 30 items (range=0-30). Higher scores mean a better outcome.
Differences between groups in scores of selective attention, inhibition, and processing speed | Before the intervention and 12 weeks later
  Selective attention, inhibition, and processing speed are measured with the Stroop Color and Word Test. Participants are asked to name the color of a series of color patches (Stroop Color Naming), read a series of color words (Stroop Word Reading), and name the color of a series of color words where the word and color do not match (e.g., the word "red" written in blue ink), Stroop Color-Word Interference. Higher scores mean a better outcome.
Differences between groups in scores of Visual scanning and processing speed | Before the intervention and 12 weeks later
  Visual scanning and processing speed are measured with the Trail-Making Test-A version. Participants are asked to connect a series of numbered circles on a page in numerical order. Higher scores mean a better outcome.
Differences between groups in scores of Executive functioning and cognitive flexibility | Before the intervention and 12 weeks later
  Executive functioning and cognitive flexibility are measured with the Trail-Making Test-B version. Participants are asked to connect a series of circles that contain both numbers and letters in alternating numerical and alphabetical order. Higher scores mean a better outcome.
Differences between groups in scores of auditory attention | Before the intervention and 12 weeks later
  Auditory attention is measured with Digit Span Forward from WAIS-IV. Participants are asked to repeat numbers in the same order as read aloud by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of working memory | Before the intervention and 12 weeks later
  Working memory is measured with Digit Span Backward from WAIS-IV. Participants are asked to repeat the numbers in the reverse order of that presented by the examiner. Higher scores mean a better outcome.
Differences between groups in scores of sustained attention and impulsivity | Before the intervention and 12 weeks later
  Conners Continuous Performance Test - 2nd edition (CPT-II) is task-oriented computerised assessment of attention-related problems. Participants are presented with a repetitive array of visual stimuli on a computer screen for 14 min. Participants are instructed to press the space bar every time a letter other than "X" appears and to not press the space bar when "X" appears. The rate of stimulus presentation varies according to 1, 2, and 4 s intervals throughout the task. Measures: Correct Detection (Higher rates indicate better outcome), Reaction times (Lower scores indicate better outcome), Omission errors (Lower rates indicate better outcome), and Commission errors (Lower rates indicate better outcome).
Differences between groups in scores of processing speed | Before the intervention and 12 weeks later
  The Digit Symbol Coding subtest from the WAIS-III is a neuropsychological assessment instrument for the detection of brain dysfunction in children and adults. It consists of replacing symbols that lack verbal meaning with numbers based on a key. Higher scores indicate better outcomes.
Differences between groups in scores of verbal memory and learning | Before the intervention and 12 weeks later
  Verbal memory and learning are measured with the Rey Auditory Verbal Learning Test (RAVLT). It is a word-learning test where five presentations of a 15-word list are given, each followed by an attempted recall. This is followed by a second 15-word interference list (list B), followed by a recall of list A. Delayed recall and recognition are also tested. Higher scores mean a better outcome.
Differences between groups in scores of phonetic fluency | Before the intervention and 12 weeks later
  Phonetic fluency is measured with the FAS test. It consists of saying words that start with a certain letter, as many words as possible must be mentioned during a specific time of 1 minute. The standard administration of the test provides three letters, the most used are the letters F, A, and S. Higher scores indicate better performance.
Differences between groups in scores of semantic verbal fluency | Before the intervention and 12 weeks later
  Semantic verbal fluency is measured with the ANIMAL test. It consists of generating the name of as many species of animals as possible within 1min. Higher scores indicate better performance.
Differences between groups in scores of memory and everyday forgetfulness | Before the intervention and 12 weeks later
  Memory and everyday forgetfulness are measured with The Memory Failures of Everyday-MFE Questionnaire is a self-reported test that allows an assessment of memory and everyday forgetfulness. It is a unifactorial questionnaire and consists of 30 items. The total score results from the sum of the scores in each item, from 1 to 30. The MFE can assess the current situation of the patients and their evolution long-term or changes due to treatment. Scores <8 represent an optimal memory function. Lower scores indicate better outcomes.
Differences between groups in word knowledge and verbal concept | Before the intervention and 12 weeks later
  Word Knowledge and verbal concept are measures with the Vocabulary subtest of The Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV). It requires the participant to try to define up to 30 words, with higher scores indicating better outcomes.
Differences between groups in self-reported executive functioning | Before the intervention and 12 weeks later
  Self-reported executive functioning is measured with The Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A), which has 75 items within nine non-overlapping theoretically and empirically derived clinical scales, including Inhibit, Shift, Emotional Control, Self-Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials. Higher scores indicate wors outcomes.

SECONDARY OUTCOMES:
Differences between groups in scores of anxiety | Before the intervention and 12 weeks later
  Anxiety is measured with the 7-item Generalized Anxiety Disorder Scale (GAD-7), a Likert-type scale with questions ranging from "not at all" (0 points) to "nearly every day" (3 points). The maximum score is 24. Higher scores mean a worse outcome.
Differences between groups in scores of depression | Before the intervention and 12 weeks later
  Depression is measured with the Patient Health Questionnaire-9 (PHQ-9) which scores each of the 9 DSM-IV criteria as "not at all" (0 points) to "nearly every day" (3 points). Higher scores mean a worse outcome.
Differences between groups in scores of Fatigue | Before the intervention and 12 weeks later
  Fatigue is measured with the Chalder Fatigue Scale, an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales. Seven items represent physical fatigue (items 1-7) and 4 represent mental fatigue (items 8-11). Each item " less than usual" (0) to " much more than usual" (3). The ratings of items are added together to calculate the total score (range=0-33). High scores represent high levels of fatigue.
Differences between groups in scores of Quality of Life | Before the intervention and 12 weeks later
  Quality of Life is measured with EuroQol a self-completion questionnaire, which consists of five questions: covering mobility, hygiene, activities, pain, and anxiety. The descriptive system divides each of the 5 dimensions into three levels of response: the absence of a problem, some problem, and extreme problem. Lower scores indicate better outcomes. In addition, the questionnaire has a plus scale where the participants rated their health state on a scale of 0-100. In this scale, higher scores indicate better outcome.
Differences between groups in cancer-related quality of life | Before the intervention and 12 weeks later
  Quality of life scales for each type of cancer will be assessed with the EORTC Quality of Life Questionnaire for Breast Cancer EORTC QLQ-BR23. The EORTC QLQ-BR23 is a breast-specific module that comprises 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss. In this scale, higher scores indicate better outcomes.
Differences between groups in Functionality | Before the intervention and 12 weeks later
  Functionality is measured with a 12-item World Health Organization Disability Assessment Schedule-II (WHODAS-II). Patients are asked to state the level of difficulty experienced, considering how they usually do the activity. The scale scores each item as "none" (1) to "cannot do" (5). The total score is calculated with an SPSS syntax, and the range varies from 0 to 100, with higher scores reflecting more significant disability.
Differences between groups in scores of Sleep Quality | Before the intervention and 12 weeks later
  Sleep Quality is measured with The Pittsburgh Sleep Quality Index (PSQI). This test presents 24 items, although only 19 are taken into account for the correction. This test is divided into 7 dimensions, namely, sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, hypnotic drugs, and daytime dysfunction. Higher scores indicate worse sleep quality.
Differences between groups in scores of performed physical activity | Before the intervention and 12 weeks later
  Performed physical activity is measured with The International Physical Activity Questionnaire (IPAQ) is a questionnaire composed of 7 questionsin order to assessthe frequency, duration, and intensity (vigorous or moderate) of the performed physical activity, walking, and sitting time during a business day for the last 7 days. Later, from the minutes obtained from the participant's answers, the METS (metabolic equivalent tasks) conversion is performed, allowing a classification, depending on the energy consumption obtained for each activity, into three categories (low, medium, high). Higher score indicate better outcome.
Differences between groups in scores of loneliness | Before the intervention and 12 weeks later
  Loneliness levels are measured through the UCLA Loneliness Scale, a widely recognized tool for measuring subjective feelings of loneliness or social isolation. The most recent version, contains 20 items rated on a scale from 1 (Never) to 4 (Always). Higher scores indicate worse outcomes.
Differences between groups in scores of psychological coping responses for cancer | Before the intervention and 12 weeks later
  Coping strategies for cancer are measured through the Mental Adjustment to Cancer Scale, a widely recognized tool for measuring subjective coping strategies that cancer patients may display. The scale has 29 items and a higher scores indicate worse outcomes.
Differences between groups in scores of fear of cancer recurrence | Before the intervention and 12 weeks later
  Fear of cancer recurrence levels are measured through the Fear of Cancer Recurrence Inventory (FCRI), a 42-item scale that is recognized as one of the psychometrically strongest measures of fear of cancer recurrence. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Spain

IPD SHARING:
Plan to Share IPD: No